CLINICAL TRIAL: NCT06085976
Title: Efficacy and Safety of Octreotide in Laparoscopic Hepatectomy Surgery: Effect on Blood Loss, Need for Vasoactive Drugs, Transfusion Requirements.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HEPA-OCT
Record Dates: First submitted 2023-09-19; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-07

CONDITIONS: Hepatic Carcinoma; Hepatic Metastasis
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Octreotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (octreotide) (Experimental): This patient will receive the treatment: Octreotide charge 100 mcgr + continuous infusion during the surgery 25 mcgr/h
  Interventions: Drug: Octreotide
- Placebo arm (saline solution) (Experimental): This patient will receive physiologic saline solution at the same infusion
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Octreotide — A loading dose of 100 mcgr of octreotide will be administered in the intervention group, diluted in 100 ml of SSF to be passed in 30 minutes.
  Subsequently, it will be administered in continuous perfusion at 25 mcgr/h in the intervention group.
  The drug can be administered through a peripheral or central venous line at the choice of the anesthesiologist, since the drug has a density that allows its administration by both routes.
  Other Names: Placebo
  Arms: Treatment arm (octreotide)
Other: Placebo — In the case of the control group, 100 ml of SSF will be administered to be passed in half an hour and then an perfusion of SSF.
  Arms: Placebo arm (saline solution)

SUMMARY:
The goal of this double-blind clinical trial is to compare the efficacy of octreotide versus placebo in laparoscopic hepatectomy surgery in patients diagnosed with resectable hepatocarcinoma or liver metastases.

The main questions it aims to answer are:

* Decrease in intraoperative bleeding measured in ml of blood lost.
* Decrease in the need for blood transfusion and use of intraoperative vasoactive drugs.

Participants will receive octreotide or placebo after signing the informed consent form.

DETAILED DESCRIPTION:
The drug will be administered during surgery, after anesthetic induction, and will be withdrawn at the end of surgery before leaving the operating room.

The patient will not receive any visit or require the performance of any other additional tests that are performed in the usual clinical practice. The monthly follow-up will coincide with the medical check-up and control analytical data will be taken. Subsequently, an attempt will be made to contact with the patient 3 months after surgery.

The duration of participation of each participant in the trial will therefore be about 3 months after surgery.

The intervention group will receive a loading dose of octreotide (100 mcgr) diluted in 100 ml of SSF to be given in half an hour and after that a continuous perfusion of 25 mcgr/h will be started until the end of the surgery.

The pharmaceutical form to be used is Sandostatin.

The control group will receive SSF as a placebo in the same sequence, first a loading dose in half an hour and then a continuous infusion of 25 mcgr/h until the end of surgery.

and then a continuous infusion until the end of the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hepatic lesions who are going to undergo hepatectomy via laparoscopy.
* The patient must be between 18 and 80 years old.
* The patient, or his/her representative, has given his/her consent to participate in the study.
* The patient must, in the opinion of the investigator, be able to comply with all the requirements of the clinical trial.
* The patient must not be allergic to the drug.

Exclusion Criteria:

* History of hypersensitivity to the drug to be administered.
* Children under 18 years of age.
* Urgent intervention.
* Intervention performed in an open manner (not laparoscopic).
* Patient's refusal to participate in the study.
* Contraindication to receive octreotide.
* Women of childbearing age (those women who are in the period between menarche and menopause). Having to present a negative pregnancy test to take part in the study.
* Pregnant or lactating women, given the absence of studies of this drug in this patient profile.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2025-08-14 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence on intraoperative bleeding. | During the time the surgery lasts.
  Decrease in intraoperative bleeding measured in ml of blood lost during laparoscopic liver resection surgery via laparoscopy.

SECONDARY OUTCOMES:
Rate of intraoperative hemodynamic stability. | During the time the surgery lasts.
  Intraoperative hemodynamic stability through haemodynamics variables.
Incidence of intraoperative transfusion. | During the time the surgery lasts.
  Decrease in transfusion during surgery due to bleeding versus placebo
Number of patients with vasoactive use. | During the time the surgery lasts.
  Decrease in use of vasoactive drugs due to hemodynamic instability versus placebo
Incidence on the improvement of hepatic function | Up to 90 days
  Observe the effects on postoperative liver function, reduction of liver enzymes.
Rate of postoperative complications | Up to 90 days
  Observe the effects on postoperative complications versus placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Universidad de Navarra, Pamplona, Spain

REFERENCES:
- [Background] Huaringa-Marcelo J, Huaman MR, Branez-Condorena A, Villacorta-Landeo P, Pinto-Ruiz DF, Urday-Ipanaque D, Garcia-Gomero D, Montes-Teves P, Lozano Miranda A. Vasoactive Agents for the Management of Acute Variceal Bleeding: A Systematic Review and Meta-analysis. J Gastrointestin Liver Dis. 2021 Mar 13;30(1):110-121. doi: 10.15403/jgld-3191. PMID 33723542
- [Background] Condron ME, Pommier SJ, Pommier RF. Continuous infusion of octreotide combined with perioperative octreotide bolus does not prevent intraoperative carcinoid crisis. Surgery. 2016 Jan;159(1):358-65. doi: 10.1016/j.surg.2015.05.036. Epub 2015 Oct 23. PMID 26603846
- [Background] Lu SC, Meng FK, Ding HG, Zhang JG, Ding L, Wang SZ. [Effects of two different dosages of octreotide on portal pressure and hepatic hemodynamics in cirrhotic portal hypertensive patients after portal-azygous devascularization and splenectomy]. Zhonghua Nei Ke Za Zhi. 2007 Apr;46(4):290-3. Chinese. PMID 17637266
- [Background] Weingarten TN, Abel MD, Connolly HM, Schroeder DR, Schaff HV. Intraoperative management of patients with carcinoid heart disease having valvular surgery: a review of one hundred consecutive cases. Anesth Analg. 2007 Nov;105(5):1192-9, table of contents. doi: 10.1213/01.ane.0000284704.57806.0b. PMID 17959940
- [Background] Woltering EA, Wright AE, Stevens MA, Wang YZ, Boudreaux JP, Mamikunian G, Riopelle JM, Kaye AD. Development of effective prophylaxis against intraoperative carcinoid crisis. J Clin Anesth. 2016 Aug;32:189-93. doi: 10.1016/j.jclinane.2016.03.008. Epub 2016 Apr 20. PMID 27290972
- [Background] Dahaba AA, Mueller G, Mattiassich G, Rumpold-Seitlinger G, Bornemann H, Rehak PH, Linck G, Mischinger HJ, Metzler H. Effect of somatostatin analogue octreotide on pain relief after major abdominal surgery. Eur J Pain. 2009 Sep;13(8):861-4. doi: 10.1016/j.ejpain.2008.10.006. Epub 2008 Dec 11. PMID 19084439
- [Background] Suc B, Msika S, Piccinini M, Fourtanier G, Hay JM, Flamant Y, Fingerhut A, Fagniez PL, Chipponi J; French Associations for Surgical Research. Octreotide in the prevention of intra-abdominal complications following elective pancreatic resection: a prospective, multicenter randomized controlled trial. Arch Surg. 2004 Mar;139(3):288-94; discussion 295. doi: 10.1001/archsurg.139.3.288. PMID 15006886
- [Background] Latchana N, Hirpara DH, Hallet J, Karanicolas PJ. Red blood cell transfusion in liver resection. Langenbecks Arch Surg. 2019 Feb;404(1):1-9. doi: 10.1007/s00423-018-1746-2. Epub 2019 Jan 3. PMID 30607533
- [Background] Hallet J, Tsang M, Cheng ES, Habashi R, Kulyk I, Hanna SS, Coburn NG, Lin Y, Law CH, Karanicolas PJ. The Impact of Perioperative Red Blood Cell Transfusions on Long-Term Outcomes after Hepatectomy for Colorectal Liver Metastases. Ann Surg Oncol. 2015 Nov;22(12):4038-45. doi: 10.1245/s10434-015-4477-4. Epub 2015 Mar 10. PMID 25752895
- [Background] Wang C, Han J, Xiao L, Jin CE, Li DJ, Yang Z. Efficacy of vasopressin/terlipressin and somatostatin/octreotide for the prevention of early variceal rebleeding after the initial control of bleeding: a systematic review and meta-analysis. Hepatol Int. 2015 Jan;9(1):120-9. doi: 10.1007/s12072-014-9594-9. Epub 2014 Dec 5. PMID 25788386
- [Background] Li JJ, Chao P, Gernsheimer J, Verma R. Octreotide for Gastrointestinal Hemorrhage from Esophageal Varices. Acad Emerg Med. 2020 Apr;27(4):339-340. doi: 10.1111/acem.13901. Epub 2019 Dec 31. No abstract available. PMID 31821652
- [Background] Berreta J, Kociak D, Romero G, Balducci A, Amaya R, Argonz J. [Endoscopic versus endoscopic plus octreotide treatment for acute variceal bleeding. Benefit according to severity at admission]. Acta Gastroenterol Latinoam. 2013 Jun;43(2):89-97. Spanish. PMID 23940908
- [Background] Sung JJ, Chung SC, Yung MY, Lai CW, Lau JY, Lee YT, Leung VK, Li MK, Li AK. Prospective randomised study of effect of octreotide on rebleeding from oesophageal varices after endoscopic ligation. Lancet. 1995 Dec 23-30;346(8991-8992):1666-9. doi: 10.1016/s0140-6736(95)92840-5. PMID 8551824
- [Background] Iannone A, Principi M, Barone M, Losurdo G, Ierardi E, Di Leo A. Gastrointestinal bleeding from vascular malformations: Is octreotide effective to rescue difficult-to-treat patients? Clin Res Hepatol Gastroenterol. 2016 Sep;40(4):373-7. doi: 10.1016/j.clinre.2016.02.003. Epub 2016 Aug 29. PMID 27595456
- [Background] Fabes J, Ambler G, Shah B, Williams NR, Martin D, Davidson BR, Spiro M. Protocol for a prospective double-blind, randomised, placebo-controlled feasibility trial of octreotide infusion during liver transplantation. BMJ Open. 2021 Dec 2;11(12):e055864. doi: 10.1136/bmjopen-2021-055864. PMID 34857585
- [Background] Sahmeddini MA, Amini A, Naderi N. The effect of octreotide on urine output during orthotopic liver transplantation and early postoperative renal function; a randomized, double-blind, placebo-controlled trial. Hepat Mon. 2013 Sep 18;13(9):e12787. doi: 10.5812/hepatmon.12787. eCollection 2013. PMID 24282425
- [Background] Williams WH 3rd, Browne RC, Bui TP, Holmes AA, Thakar D. Case report on intravenous octreotide for the treatment of intraoperative vasoplegia following thymoma resection. SAGE Open Med Case Rep. 2019 Feb 8;7:2050313X19827744. doi: 10.1177/2050313X19827744. eCollection 2019. PMID 30800305
- [Background] Edelson J, Basso JE, Rockey DC. Updated strategies in the management of acute variceal haemorrhage. Curr Opin Gastroenterol. 2021 May 1;37(3):167-172. doi: 10.1097/MOG.0000000000000723. PMID 33769373
- See also: Byram, S., Gupta, R., Ander, M., Edelstein, S. & Andreatta, B. (2015). Effects of Continuous Octreotide Infusion on Intraoperative Transfusion Requirements During Orthotopic Liver Transplantation. Transplantation Proceedings, 47(9), 2712-2714. — https://doi.org/10.1016/j.transproceed.2015.07.036
- See also: El Nakeeb, A., ElGawalby, A., A. Ali, MEfficacy of octreotide in the prevention of complications after pancreaticoduodenectomy in patients with soft pancreas and non-dilated pan — https://doi.org/10.1016/j.hbpd.2018.01.015
- See also: Terlipressin and the Treatment o — https://doi.org/10.1053/j.ajkd.2021.08.016
- See also: Pisani, A., Sabbatini, M., Imbriaco, M., Riccio, E., Rubis, N., Prinster, A., Perna, A., Liuzzi, R., Spinelli, L., Santangelo, M., Remuzzi, G., Ruggenenti, P., Pisani, A., Sabbatini, M., Ruggenenti, P., Remuzzi, G., Pisani, A., Visciano, B., Amicone, M., — https://doi.org/10.1016/j.cgh.2015.12.049
- See also: Somatostatin analogue, Octreotide, improves restraint stress-induced liver injury by ameliorating oxidative stress, inflammatory response, and activation of hepatic stellate cells. Cell Stress and Chaperones — https://doi.org/10.1007/s12192-018-0929-7